CLINICAL TRIAL: NCT06165965
Title: A Randomized, Open-label, Two-sequence, and Two-period Crossover Study to Evaluate the Pharmacokinetics and Safety Between the Administration of JLP-2008 and the Co-admin. of JT-001, and JT-002 for Healthy Subjects in Fasted State
Brief Title: To Evaluate the Safety and Pharmacokinetic Characteristics After the Administration of JT-001, JT-002 and JLP-2008
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JP-2008-101
Record Dates: First submitted 2023-11-22; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Healthy Adult
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment(Experimental): JLP-2008 (Experimental): - Group I(Peroid I-Comparator[JT-001,JT-002], Peroid II-JLP-2008), Group II(Period I-JLP-2008, Period II-Comparator[JT-001,JT-002])
  Interventions: Drug: SGLT2 inhibitor
- Control(Active Comparator): JC-013 (Active Comparator): - Group I(Peroid I-Comparator[JT-001,JT-002], Peroid II-JLP-2008), Group II(Period I-JLP-2008, Period II-Comparator[JT-001,JT-002])
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — SGLT2 dual inhibitor

SUMMARY:
To evaluate the safety and pharmacokinetic characteristics after the administration of JT-001, JT-002 and JLP-2008

DETAILED DESCRIPTION:
A randomized, open-label, single oral dosing, two-sequence, and two-period crossover study to evaluate the pharmacokinetics and safety between the administration of JLP-2008 and the co-administration of JT-001, and JT-002 for healthy subjects in fasted state

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between 19 and 55 years of age at the time of screening test
2. At the time of the screening test, a subject weighing more than 50 kg for men and 45 kg for women, and a body mass index (BMI) of 18.0 kg/m2 or more and 30.0 kg/m2 or less.
3. After receiving a detailed explanation of this clinical trial and fully understanding it, those who voluntarily decide to participate and give written consent before the screening procedure

Exclusion Criteria:

1. Those with a clinically significant history of hypersensitivity, intolerance, or anaphylaxis to the main ingredient or other components of the investigational product
2. Those who have clinically siginificant medical history of liver (severe liver disorders, etc.), kidneys (severe renal disorders, etc.), digestive system (pancreatitis, etc.), respiratory system, musculoskeletal system, endocrine system (diabetic ketoacidosis, diabetic coma and precoma, type 1 Diabetes mellitus), neuropsychiatric, hematologic/oncological, and cardiovascular (heart failure, orthostatic hypotension, etc.)
3. Those with a history of Gastrointestinal disease (e.g. Crohn's disease, ulcerative disease, etc.) or surgery (excluding appendectomy, hernia surgery, endoscopic polyp surgery, hemorrhoids, dentition, and fistula surgery) that may affect the absorption of the investigational product
4. Persons judged to be unsuitable as trial subjects in the test items conducted during screening

   * Blood ALT, AST, Total bilirubin > 2 times the upper limit of normal range
   * eGFR < 60 mL/min/1.73m2 (using CKD-EPI formula)
   * HBsAg, HCV Ab, HIV, Syphilis regain test (RPR) results are positive
   * Vital signs measured in the sitting position after resting for more than 3 minutes: systolic blood pressure > 160 mmHg or < 90 mmHg, or diastolic blood pressure > 100 mmHg or < 50 mmHg

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
AUC over24H of JLP-2008 | 24 hours
Cmax of JLP-2008 | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Bundang CHA university global clinical trials center Institutional Review Board, Gyeonggi-do, Bundang-gu, South Korea